CLINICAL TRIAL: NCT04736056
Title: Mindfulness and Cognitive Behavioral Therapy for Sleep in Cancer
Brief Title: Mindfulness and CBT for Sleep
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00107338
Record Dates: First submitted 2021-01-29; First posted 2021-02-03 (Actual); Results first posted 2024-12-02 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-10

CONDITIONS: Hematologic Malignancy
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Intervention Model Description: Single Group Assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Mindfulness-Based Therapy for Insomnia with Cognitive-Behavioral Symptom Coping Skills (Experimental): Mindfulness-Based Therapy for Insomnia with Cognitive-Behavioral Symptom Coping Skills (MBTI+)
  The MBTI+ intervention will train participants in mindfulness-based sleep strategies and behavioral symptom management techniques. The MBTI+ intervention will consist of 6 weekly sessions that will last between 60 and 75 minutes.
  Interventions: Behavioral: Mindfulness-Based Therapy for Insomnia with Cognitive-Behavioral Symptom Coping Skills

INTERVENTIONS:
Behavioral: Mindfulness-Based Therapy for Insomnia with Cognitive-Behavioral Symptom Coping Skills — Mindfulness-based sleep strategies and cognitive-behavioral symptom coping skills.

SUMMARY:
Patients with hematologic cancer frequently report significant difficulties with sleep in the months after discharge from inpatient chemotherapy. Poor sleep quality can contribute to and perpetuate problems with daytime fatigue, pain, and distress that are common among patients with hematologic cancer. There is a need for behavioral interventions that address insomnia and daytime fatigue, pain, and distress once hematologic cancer patients have returned home after inpatient chemotherapy. Mindfulness-Based Therapy for Insomnia (MBTI) is a new approach to treating insomnia. This group-based intervention combines sleep restriction and stimulus control with mindfulness principles and exercises to reduce worry and promote positive responses to insomnia. To date, MBTI has not been applied to patients with hematologic cancer. If MBTI is to meet the needs of hematologic cancer patients, it must be adapted in several ways. First, because hematologic cancer patients are immunosuppressed, MBTI needs to be adapted for one-to-one delivery. Second, because hematologic cancer patients experience significant daytime fatigue, pain, and distress, MBTI needs to be adapted to include systematic training in coping skills for these symptoms. The investigators propose to develop and pilot test an adapted MBTI (MBTI+) protocol for hematologic cancer patients reporting insomnia, fatigue, pain, and/or distress after inpatient chemotherapy. The study will be conducted in two phases. In Phase I, the study team will use focus groups with hematologic cancer patients and hematology-oncology providers to guide development along with user testing with hematologic cancer patients reporting insomnia and daytime symptoms of fatigue, pain, and/or distress. Phase II will involve a small single-arm pilot to examine the feasibility, acceptability, and examine pre- to post-intervention primary (insomnia) and secondary (fatigue, pain, distress, mindfulness, self-efficacy) outcomes of the MBTI+ protocol. MBTI+ will consist of six, 60- to 75-minute therapy sessions delivered either in-person or via videoconferencing technology. Study measures will be collected at baseline, immediately post-intervention, and 1-month post-intervention.

ELIGIBILITY:
Inclusion Criteria:

* an initial or recurrent diagnosis of hematologic malignancy
* within 8 weeks of discharge home after inpatient chemotherapy or CAR-T therapy
* total score of 8 or greater on the Insomnia Severity Index (ISI)
* score of 5 or greater on the MD Anderson Symptom Inventory Scale for "worst" fatigue, pain, or distress, and report that these symptoms interfered with at least two activities of living (i.e., general activity, mood, work) in the last week at 3 or greater on a 0="Did not interfere" to 10="Interfered completely" scale
* ability to speak and read English, and hearing and vision that allows for completion of sessions and assessments

Exclusion Criteria:

* reported or suspected cognitive impairment subsequently informed by a Folstein Mini-Mental Status Examination of <25
* presence of a serious psychiatric (e.g., schizophrenia, suicidal intent) or medical condition (e.g., seizure disorder, narcolepsy) indicated by medical chart, treating oncologist or other medical provider that would contraindicate safe participation
* expected survival of 6 months or less

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2023-05-19 (Actual); Study Completion 2023-05-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tamara J Somers, PhD, Principal Investigator — Duke University
Locations (1):
- Duke Cancer Institute, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fisher HM, Hyland KA, Miller SN, Amaden GH, Diachina A, Ulmer CS, Danforth M, LeBlanc TW, Somers TJ, Keefe FJ. Mindful Night-to-Day: A Pilot Feasibility Trial of a Mindfulness-Based Insomnia and Symptom Management Intervention for Patients with Hematologic Cancer. Behav Sleep Med. 2024 Sep-Oct;22(5):674-696. doi: 10.1080/15402002.2024.2339819. Epub 2024 Apr 10. PMID 38597262

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase 1 Part 1: Focus Group Patients (Months 0-6): Patients with hematologic cancer endorsing insomnia symptoms, and symptoms of fatigue, pain, and/or distress. Patients completed a one-time, 60-minute, telehealth focus group to share about their symptoms and impressions of the proposed intervention protocol.
- Phase 1 Part 1: Focus Group Providers (Months 0-6): Hematology-oncology providers caring for patients with hematologic cancer. Providers completed a one-time, 60-minute, telehealth focus group to share about common hematologic cancer symptoms and their impressions of the proposed intervention protocol.
- Phase 1 Part 2: Patient User Testing (Months 6-12): Patients with hematologic cancer endorsing insomnia symptoms, and symptoms of fatigue, pain, and/or distress participated in user testing of the proposed intervention protocol prior to the single-arm pilot.
  Intervention:
  Mindfulness-Based Therapy for Insomnia with Cognitive-Behavioral Symptom Coping Skills (MBTI+)
  The MBTI+ intervention will train participants in mindfulness-based sleep strategies and behavioral symptom management techniques. The MBTI+ intervention will consist of 6 weekly sessions that will last between 60 and 75 minutes.
  Mindfulness-Based Therapy for Insomnia with Cognitive-Behavioral Symptom Coping Skills: Mindfulness-based sleep strategies and cognitive-behavioral symptom coping skills.
- Phase 2: Single-Arm Pilot (Months 12-23): Patients with hematologic cancer endorsing insomnia symptoms, and symptoms of fatigue, pain, and/or distress participated in a single-arm pilot trial.
  Intervention: Mindfulness-Based Therapy for Insomnia with Cognitive-Behavioral Symptom Coping Skills (MBTI+)
  The MBTI+ intervention will train participants in mindfulness-based sleep strategies and behavioral symptom management techniques. The MBTI+ intervention will consist of 6 weekly sessions that will last between 60 and 75 minutes.
  Mindfulness-Based Therapy for Insomnia with Cognitive-Behavioral Symptom Coping Skills: Mindfulness-based sleep strategies and cognitive-behavioral symptom coping skills.
  Mindfulness-Based Therapy for Insomnia with Cognitive-Behavioral Symptom Coping Skills: Mindfulness-based sleep strategies and cognitive-behavioral symptom coping skills.
Period: Overall Study
Arm/Group | Phase 1 Part 1: Focus Group Patients (Months 0-6) | Phase 1 Part 1: Focus Group Providers (Months 0-6) | Phase 1 Part 2: Patient User Testing (Months 6-12) | Phase 2: Single-Arm Pilot (Months 12-23)
Started | 14 | 6 | 5 | 32
Completed | 10 | 6 | 3 | 30
Not Completed | 4 | 0 | 2 | 2
Not completed — Death | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 1 | 0 | 1 | 1
Not completed — Withdrawal by Subject | 2 | 0 | 0 | 0
Not completed — Physician Decision | 1 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Phase 2: Single-Arm Pilot (Months 12-23): Patients with hematologic cancer endorsing insomnia symptoms, and symptoms of fatigue, pain, and/or distress participated in a single-arm pilot trial.
  Intervention: Mindfulness-Based Therapy for Insomnia with Cognitive-Behavioral Symptom Coping Skills (MBTI+)
  The MBTI+ intervention will train participants in mindfulness-based sleep strategies and behavioral symptom management techniques. The MBTI+ intervention will consist of 6 weekly sessions that will last between 60 and 75 minutes.
  Mindfulness-Based Therapy for Insomnia with Cognitive-Behavioral Symptom Coping Skills: Mindfulness-based sleep strategies and cognitive-behavioral symptom coping skills.
- Total: Total of all reporting groups
Arm/Group | Phase 1 Part 1: Focus Group Patients (Months 0-6) | Phase 1 Part 1: Focus Group Providers (Months 0-6) | Phase 1 Part 2: Patient User Testing (Months 6-12) | Phase 2: Single-Arm Pilot (Months 12-23) | Total
Number analyzed (Participants) | 14 | 6 | 5 | 32 | 57
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.86 (15.85) | 36.00 (10.83) | 36.00 (12.27) | 50.75 (19.64) | 49.39 (17.35)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 4 | 17 | 33
  Male | 8 | 0 | 1 | 15 | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 4 | 4
  Not Hispanic or Latino | 14 | 6 | 5 | 28 | 53
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 4 | 1 | 2 | 3 | 10
  White | 10 | 5 | 3 | 26 | 44
  More than one race | 0 | 0 | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 14 | 6 | 5 | 32 | 57

OUTCOME MEASURES:

1. Primary Outcome: Feasibility as Measured by Number of Participants Accrued to Single-arm Pilot
Description: Treatment feasibility will be indicated by meeting target study accrual (i.e., 30 participants consented and enrolled for single-arm pilot).
Time Frame: 12 weeks (post-intervention)
Population: Individuals who completed phone screening. Only applicable to Phase 2 participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2: Single-Arm Pilot (Months 12-23)
Number analyzed (Participants) | 79
Participants | 32

2. Primary Outcome: Feasibility as Measured by Study Attrition at Post-intervention Follow-up
Description: Treatment feasibility will be indicated by less than or equal to 20% study attrition at post-intervention follow-up.
Time Frame: 12 weeks (post-intervention)
Population: Participants consented and enrolled to complete the intervention (i.e., user testing and single-arm pilot participants).
Measure: Number; unit: percentage of attrition
Groups:
- Phase 1 Part 2: Patient User Testing (Months 6-12) and Phase 2: Single-Arm Pilot (Months 12-23): Patients with hematologic cancer endorsing insomnia symptoms, and symptoms of fatigue, pain, and/or distress that consented and enrolled to complete the intervention protocol (i.e., user testing and the single-arm pilot).
  Intervention:
  Mindfulness-Based Therapy for Insomnia with Cognitive-Behavioral Symptom Coping Skills (MBTI+)
  The MBTI+ intervention will train participants in mindfulness-based sleep strategies and behavioral symptom management techniques. The MBTI+ intervention will consist of 6 weekly sessions that will last between 60 and 75 minutes.
  Mindfulness-Based Therapy for Insomnia with Cognitive-Behavioral Symptom Coping Skills: Mindfulness-based sleep strategies and cognitive-behavioral symptom coping skills.
Arm/Group | Phase 1 Part 2: Patient User Testing (Months 6-12) and Phase 2: Single-Arm Pilot (Months 12-23)
Number analyzed (Participants) | 37
percentage of attrition | 8.10

3. Primary Outcome: Feasibility as Measured by Adherence to the Intervention
Description: Adherence will be indicated by at least 80% of the participants completing all 6 intervention sessions.
Time Frame: 12 weeks (post-intervention)
Population: Participants consented and enrolled to complete the intervention (i.e., user testing and single-arm pilot participants).
Measure: Number; unit: percentage of participants
Arm/Group | Phase 1 Part 2: Patient User Testing (Months 6-12) and Phase 2: Single-Arm Pilot (Months 12-23)
Number analyzed (Participants) | 37
percentage of participants | 83.80

4. Primary Outcome: Acceptability as Measured by the Client Satisfaction Questionnaire (CSQ)
Description: Acceptability will be indicated by at least 80% of participants who completed the intervention protocol reporting satisfaction with the protocol on the CSQ (i.e., mean of at least 3 out of 4). The CSQ is a 10 item self-report measure with item responses ranging from 1 to 4, with higher scores indicating greater satisfaction. All 10 items were averaged to obtain a mean score (range: 1 - 4). The number of participants with a mean CSQ score of at least 3 out of 4 was tabulated and then converted to a percentage of patients.
Time Frame: 12 weeks (post-intervention)
Population: Participants consented and enrolled to complete the intervention (i.e., user testing and single-arm pilot participants) who completed the intervention protocol.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1 Part 2: Patient User Testing (Months 6-12) and Phase 2: Single-Arm Pilot (Months 12-23)
Number analyzed (Participants) | 31
Participants | 29

5. Primary Outcome: Insomnia Symptoms as Measured by the Insomnia Symptom Index (ISI)
Description: Insomnia symptoms will be measured using the 7-item Insomnia Symptom Index (ISI). Scores on the ISI range from 0 to 28 with higher scores indicating more severe insomnia symptoms.
Time Frame: 0 weeks, 12 weeks, 16 weeks (baseline, post-intervention, 4-weeks post-intervention)
Population: Participants that consented and enrolled to complete the intervention (i.e., user testing and single-arm pilot participants).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Phase 1 Part 2: Patient User Testing (Months 6-12) and Phase 2: Single-Arm Pilot (Months 12-23)
Number analyzed (Participants) | 37
score on a scale
  0 weeks | 13.45 (6.19)
  12 weeks | 6.26 (4.46)
  16 weeks | 6.07 (3.99)
Statistical Analysis 1: Comparison: Phase 1 Part 2: Patient User Testing (Months 6-12) and Phase 2: Single-Arm Pilot (Months 12-23); 0 to 12 weeks; Test type: Other; Cohen's d effect size = 1.20, 95% CI 2-sided [0.73 to 1.66]
Statistical Analysis 2: Comparison: Phase 1 Part 2: Patient User Testing (Months 6-12) and Phase 2: Single-Arm Pilot (Months 12-23); 0 to 16 weeks; Test type: Other; Cohen's d effect size = 1.07, 95% CI 2-sided [0.61 to 1.51]

6. Secondary Outcome: Fatigue Severity as Measured by the Fatigue Symptom Inventory (FSI)
Description: Fatigue symptoms will be assessed using the 11-item Fatigue Symptom Inventory (FSI). Four items measure fatigue severity. Seven items measure fatigue interference. Scores on the FSI for fatigue severity and interference range from 0 to 10 with higher scores indicating higher fatigue severity and interference.
Time Frame: 0 weeks, 12 weeks, 16 weeks (baseline, post-intervention, 4-weeks post-intervention)
Population: Participants consented and enrolled to complete the intervention (i.e., user testing and single-arm pilot participants).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Phase 1 Part 2: Patient User Testing (Months 6-12) and Phase 2: Single-Arm Pilot (Months 12-23)
Number analyzed (Participants) | 37
score on a scale
  0 weeks | 4.48 (1.97)
  12 weeks | 3.69 (2.03)
  16 weeks | 4.06 (2.32)
Statistical Analysis 1: Comparison: Phase 1 Part 2: Patient User Testing (Months 6-12) and Phase 2: Single-Arm Pilot (Months 12-23); 0 to 12 weeks; Test type: Other; Cohen's d effect size = 0.35, 95% CI 2-sided [-0.02 to 0.71]
Statistical Analysis 2: Comparison: Phase 1 Part 2: Patient User Testing (Months 6-12) and Phase 2: Single-Arm Pilot (Months 12-23); 0 to 16 weeks; Test type: Other; Cohen's d effect size = 0.25, 95% CI 2-sided [-0.12 to 0.61]

7. Secondary Outcome: Fatigue Interference as Measured by the Fatigue Symptom Inventory (FSI)
Description: as for outcome 6
Time Frame: 0 weeks, 12 weeks, 16 weeks (baseline, post-intervention, 4-weeks post-intervention)
Population: Participants consented and enrolled to complete the intervention (i.e., user testing and single-arm pilot participants).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Phase 1 Part 2: Patient User Testing (Months 6-12) and Phase 2: Single-Arm Pilot (Months 12-23)
Number analyzed (Participants) | 37
score on a scale
  0 weeks | 4.18 (2.49)
  12 weeks | 2.70 (2.55)
  16 weeks | 3.09 (2.44)
Statistical Analysis 1: Comparison: Phase 1 Part 2: Patient User Testing (Months 6-12) and Phase 2: Single-Arm Pilot (Months 12-23); 0 to 12 weeks; Test type: Other; Cohen's d effect size = 0.78, 95% CI 2-sided [0.38 to 1.18]
Statistical Analysis 2: Comparison: Phase 1 Part 2: Patient User Testing (Months 6-12) and Phase 2: Single-Arm Pilot (Months 12-23); 0 to 16 weeks; Test type: Other; Cohen's d effect size = 0.50, 95% CI 2-sided [0.11 to 0.87]

8. Secondary Outcome: Pain Severity as Measured by the Brief Pain Inventory-Short Form (BPI-SF)
Description: Pain symptoms will be measured using the 11-item Brief Pain Inventory-Short Form (BPI-SF). Four items measure pain severity. Scores on the BPI-SF for pain severity range from 0 to 10 with higher scores indicating higher pain severity.
Time Frame: 0 weeks, 12 weeks, 16 weeks (baseline, post-intervention, 4-weeks post-intervention)
Population: Participants consented and enrolled to complete the intervention (i.e., user testing and single-arm pilot participants).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Phase 1 Part 2: Patient User Testing (Months 6-12) and Phase 2: Single-Arm Pilot (Months 12-23)
Number analyzed (Participants) | 37
score on a scale
  0 weeks | 2.59 (2.19)
  12 weeks | 2.13 (2.01)
  16 weeks | 1.79 (1.89)
Statistical Analysis 1: Comparison: Phase 1 Part 2: Patient User Testing (Months 6-12) and Phase 2: Single-Arm Pilot (Months 12-23); 0 to 12 weeks; Test type: Other; Cohen's d effect size = 0.23, 95% CI 2-sided [-0.13 to 0.58]
Statistical Analysis 2: Comparison: Phase 1 Part 2: Patient User Testing (Months 6-12) and Phase 2: Single-Arm Pilot (Months 12-23); 0 to 16 weeks; Test type: Other; Cohen's d effect size = 0.31, 95% CI 2-sided [-0.05 to 0.68]

9. Secondary Outcome: Pain Interference as Measured by the Brief Pain Inventory-Short Form (BPI-SF)
Description: Pain symptoms will be measured using the 11-item Brief Pain Inventory-Short Form (BPI-SF). Seven items measure pain interference. Scores on the BPI-SF for pain interference range from 0 to 10 with higher scores indicating higher pain interference.
Time Frame: 0 weeks, 12 weeks, 16 weeks (baseline, post-intervention, 4-weeks post-intervention)
Population: Participants consented and enrolled to complete the intervention (i.e., user testing and single-arm pilot participants).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Phase 1 Part 2: Patient User Testing (Months 6-12) and Phase 2: Single-Arm Pilot (Months 12-23)
Number analyzed (Participants) | 37
score on a scale
  0 weeks | 3.35 (3.18)
  12 weeks | 2.57 (2.87)
  16 weeks | 1.85 (2.26)
Statistical Analysis 1: Comparison: Phase 1 Part 2: Patient User Testing (Months 6-12) and Phase 2: Single-Arm Pilot (Months 12-23); 0 to 12 weeks; Test type: Other; Cohen's d effect size = 0.32, 95% CI 2-sided [-0.04 to 0.68]
Statistical Analysis 2: Comparison: Phase 1 Part 2: Patient User Testing (Months 6-12) and Phase 2: Single-Arm Pilot (Months 12-23); 0 to 16 weeks; Test type: Other; Cohen's d effect size = 0.61, 95% CI 2-sided [0.22 to 1.00]

10. Secondary Outcome: Severity of Anxiety Symptoms as Measured by the Hospital Anxiety and Depression Scale (HADS)
Description: Anxiety symptoms will be measured using the 14-item Hospital Anxiety and Depression Scale (HADS). Seven items measure severity of anxiety symptoms. Scores for anxiety symptom severity range from 0 to 21 with higher scores indicating more severe anxiety.
Time Frame: 0 weeks, 12 weeks, 16 weeks (baseline, post-intervention, 4-weeks post-intervention)
Population: Participants consented and enrolled to complete the intervention (i.e., user testing and single-arm pilot participants).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Phase 1 Part 2: Patient User Testing (Months 6-12) and Phase 2: Single-Arm Pilot (Months 12-23)
Number analyzed (Participants) | 37
score on a scale
  0 weeks | 6.65 (4.22)
  12 weeks | 5.55 (4.08)
  16 weeks | 5.47 (4.33)
Statistical Analysis 1: Comparison: Phase 1 Part 2: Patient User Testing (Months 6-12) and Phase 2: Single-Arm Pilot (Months 12-23); 0 to 12 weeks; Test type: Other; Cohen's d effect size = 0.38, 95% CI 2-sided [0.01 to 0.74]
Statistical Analysis 2: Comparison: Phase 1 Part 2: Patient User Testing (Months 6-12) and Phase 2: Single-Arm Pilot (Months 12-23); 0 to 16 weeks; Test type: Other; Cohen's d effect size = 0.47, 95% CI 2-sided [0.09 to 0.85]

11. Secondary Outcome: Severity of Depressive Symptoms as Measured by the Hospital Anxiety and Depression Scale (HADS)
Description: Depressive symptoms will be measured using the 14-item Hospital Anxiety and Depression Scale (HADS). Seven items measure severity of depressive symptoms. Scores for depressive symptom severity range from 0 to 21 with higher scores indicating more severe depressive symptoms.
Time Frame: 0 weeks, 12 weeks, 16 weeks (baseline, post-intervention, 4-weeks post-intervention)
Population: Participants consented and enrolled to complete the intervention (i.e., user testing and single-arm pilot participants).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Phase 1 Part 2: Patient User Testing (Months 6-12) and Phase 2: Single-Arm Pilot (Months 12-23)
Number analyzed (Participants) | 37
score on a scale
  0 weeks | 6.61 (4.26)
  12 weeks | 5.74 (4.67)
  16 weeks | 5.20 (4.00)
Statistical Analysis 1: Comparison: Phase 1 Part 2: Patient User Testing (Months 6-12) and Phase 2: Single-Arm Pilot (Months 12-23); 0 to 12 weeks; Test type: Other; Cohen's d effect size = 0.29, 95% CI 2-sided [-0.07 to 0.65]
Statistical Analysis 2: Comparison: Phase 1 Part 2: Patient User Testing (Months 6-12) and Phase 2: Single-Arm Pilot (Months 12-23); Test type: Other; Cohen's d effect size = 0.60, 95% CI 2-sided [0.21 to 0.99]

12. Secondary Outcome: Severity of Somatic Hyperarousal Symptoms
Description: Hyperarousal symptoms will be measured using the 16-item Pre-Sleep Arousal Scale (PSAS). Eight items measure severity of somatic hyperarousal symptoms. Scores for somatic hyperarousal symptom severity range from 8 to 40 with higher scores indicating worse somatic hyperarousal severity.
Time Frame: 0 weeks, 12 weeks, 16 weeks (baseline, post-intervention, 4-weeks post-intervention)
Population: Participants consented and enrolled to complete the intervention (i.e., user testing and single-arm pilot participants).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Phase 1 Part 2: Patient User Testing (Months 6-12) and Phase 2: Single-Arm Pilot (Months 12-23)
Number analyzed (Participants) | 37
score on a scale
  0 weeks | 14.42 (5.89)
  12 weeks | 11.65 (3.08)
  16 weeks | 11.90 (3.99)
Statistical Analysis 1: Comparison: Phase 1 Part 2: Patient User Testing (Months 6-12) and Phase 2: Single-Arm Pilot (Months 12-23); 0 to 12 weeks; Test type: Other; Cohen's d effect size = 0.54, 95% CI 2-sided [0.16 to 0.91]
Statistical Analysis 2: Comparison: Phase 1 Part 2: Patient User Testing (Months 6-12) and Phase 2: Single-Arm Pilot (Months 12-23); 0 to 16 weeks; Test type: Other; Cohen's d effect size = 0.51, 95% CI 2-sided [0.12 to 0.89]

13. Secondary Outcome: Severity of Cognitive Hyperarousal Symptoms
Description: Hyperarousal symptoms will be measured using the 16-item Pre-Sleep Arousal Scale (PSAS). Eight items measure severity of cognitive hyperarousal symptoms. Scores for cognitive hyperarousal symptom severity range from 8 to 40 with higher scores indicating worse cognitive hyperarousal severity.
Time Frame: 0 weeks, 12 weeks, 16 weeks (baseline, post-intervention, 4-weeks post-intervention)
Population: Participants consented and enrolled to complete the intervention (i.e., user testing and single-arm pilot participants).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Phase 1 Part 2: Patient User Testing (Months 6-12) and Phase 2: Single-Arm Pilot (Months 12-23)
Number analyzed (Participants) | 37
score on a scale
  0 weeks | 18.61 (7.16)
  12 weeks | 15.13 (5.48)
  16 weeks | 15.40 (6.73)
Statistical Analysis 1: Comparison: Phase 1 Part 2: Patient User Testing (Months 6-12) and Phase 2: Single-Arm Pilot (Months 12-23); 0 to 12 weeks; Test type: Other; Cohen's d effect size = 0.89, 95% CI 2-sided [0.47 to 1.30]
Statistical Analysis 2: Comparison: Phase 1 Part 2: Patient User Testing (Months 6-12) and Phase 2: Single-Arm Pilot (Months 12-23); 0 to 16 weeks; Test type: Other; Cohen's d effect size = 0.66, 95% CI 2-sided [0.26 to 1.05]

14. Secondary Outcome: Mindfulness Skills as Measured by the Kentucky Inventory of Mindfulness Skills (KIMS): Observing
Description: Mindfulness skills (i.e., observing, describing, acting with awareness, and accepting/non-judgement) will be measured using the 39-item Kentucky Inventory of Mindfulness Skills (KIMS). Observing (range: 12-60) is measured by 12 items. Higher scores indicate higher levels of observing skills.
Time Frame: 0 weeks, 12 weeks, 16 weeks (baseline, post-intervention, 4-weeks post-intervention)
Population: Participants consented and enrolled to complete the intervention (i.e., user testing and single-arm pilot participants).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Phase 1 Part 2: Patient User Testing (Months 6-12) and Phase 2: Single-Arm Pilot (Months 12-23)
Number analyzed (Participants) | 37
score on a scale
  0 weeks | 36.29 (9.00)
  12 weeks | 39.23 (8.46)
  16 weeks | 39.37 (9.32)
Statistical Analysis 1: Comparison: Phase 1 Part 2: Patient User Testing (Months 6-12) and Phase 2: Single-Arm Pilot (Months 12-23); 0 to 12 weeks; Test type: Other; Cohen's d effect size = -0.40, 95% CI 2-sided [-0.76 to -0.03]
Statistical Analysis 2: Comparison: Phase 1 Part 2: Patient User Testing (Months 6-12) and Phase 2: Single-Arm Pilot (Months 12-23); 0 to 16 weeks; Test type: Other; Cohen's d effect size = -0.34, 95% CI 2-sided [-0.71 to 0.03]

15. Secondary Outcome: Mindfulness Skills as Measured by the Kentucky Inventory of Mindfulness Skills (KIMS): Describing
Description: Mindfulness skills (i.e., observing, describing, acting with awareness, and accepting/non-judgement) will be measured using the 39-item Kentucky Inventory of Mindfulness Skills (KIMS). Describing (range: 8-40) is measured by eight items. Higher scores indicate higher levels of describing skills.
Time Frame: 0 weeks, 12 weeks, 16 weeks (baseline, post-intervention, 4-weeks post-intervention)
Population: Participants consented and enrolled to complete the intervention (i.e., user testing and single-arm pilot participants).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Phase 1 Part 2: Patient User Testing (Months 6-12) and Phase 2: Single-Arm Pilot (Months 12-23)
Number analyzed (Participants) | 37
score on a scale
  0 weeks | 28.74 (5.85)
  12 weeks | 28.74 (5.68)
  16 weeks | 29.70 (5.68)
Statistical Analysis 1: Comparison: Phase 1 Part 2: Patient User Testing (Months 6-12) and Phase 2: Single-Arm Pilot (Months 12-23); 0 to 12 weeks; Test type: Other; Cohen's d effect size = 0.00, 95% CI 2-sided [-0.35 to 0.35]
Statistical Analysis 2: Comparison: Phase 1 Part 2: Patient User Testing (Months 6-12) and Phase 2: Single-Arm Pilot (Months 12-23); 0 to 16 weeks; Test type: Other; Cohen's d effect size = -0.28, 95% CI 2-sided [-0.64 to 0.09]

16. Secondary Outcome: Mindfulness Skills as Measured by the Kentucky Inventory of Mindfulness Skills (KIMS): Acting With Awareness
Description: Mindfulness skills (i.e., observing, describing, acting with awareness, and accepting/non-judgement) will be measured using the 39-item Kentucky Inventory of Mindfulness Skills (KIMS). Acting with awareness (range: 10-50) is measured by ten items. Higher scores indicate higher levels of acting with awareness skills.
Time Frame: 0 weeks, 12 weeks, 16 weeks (baseline, post-intervention, 4-weeks post-intervention)
Population: Participants consented and enrolled to complete the intervention (i.e., user testing and single-arm pilot participants).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Phase 1 Part 2: Patient User Testing (Months 6-12) and Phase 2: Single-Arm Pilot (Months 12-23)
Number analyzed (Participants) | 37
score on a scale
  0 weeks | 32.32 (5.78)
  12 weeks | 32.77 (5.52)
  16 weeks | 31.57 (5.46)
Statistical Analysis 1: Comparison: Phase 1 Part 2: Patient User Testing (Months 6-12) and Phase 2: Single-Arm Pilot (Months 12-23); Test type: Other; Cohen's d effect size = 0.10, 95% CI 2-sided [-0.45 to 0.26]
Statistical Analysis 2: Comparison: Phase 1 Part 2: Patient User Testing (Months 6-12) and Phase 2: Single-Arm Pilot (Months 12-23); 0 to 16 weeks; Test type: Other; Cohen's d effect size = 0.09, 95% CI 2-sided [-0.27 to 0.45]

17. Secondary Outcome: Mindfulness Skills as Measured by the Kentucky Inventory of Mindfulness Skills (KIMS): Accepting/Non-judgement
Description: Mindfulness skills (i.e., observing, describing, acting with awareness, and accepting/non-judgement) will be measured using the 39-item Kentucky Inventory of Mindfulness Skills (KIMS). Accepting is measured by nine items (range: 9-45). Higher scores indicate higher levels of accepting skills.
Time Frame: 0 weeks, 12 weeks, 16 weeks (baseline, post-intervention, 4-weeks post-intervention)
Population: Participants consented and enrolled to complete the intervention (i.e., user testing and single-arm pilot participants).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Phase 1 Part 2: Patient User Testing (Months 6-12) and Phase 2: Single-Arm Pilot (Months 12-23)
Number analyzed (Participants) | 37
score on a scale
  0 weeks | 32.00 (8.43)
  12 weeks | 34.29 (5.72)
  16 weeks | 33.77 (8.16)
Statistical Analysis 1: Comparison: Phase 1 Part 2: Patient User Testing (Months 6-12) and Phase 2: Single-Arm Pilot (Months 12-23); 0 to 12 weeks; Test type: Other; Cohen's d effect size = -.035, 95% CI 2-sided [-0.71 to 0.01]
Statistical Analysis 2: Comparison: Phase 1 Part 2: Patient User Testing (Months 6-12) and Phase 2: Single-Arm Pilot (Months 12-23); 0 to 16 weeks; Test type: Other; Cohen's d effect size = -0.29, 95% CI 2-sided [-0.65 to 0.08]

18. Secondary Outcome: Self-efficacy for Symptom Management as Measured by the Self-Efficacy for Management Chronic Disease Scale (SEMCD)
Description: SEMCD scores range from 0 to 10 with higher scores indicating greater self-efficacy for symptom management.
Time Frame: 0 weeks, 12 weeks, 16 weeks (baseline, post-intervention, 4-weeks post-intervention)
Population: Participants consented and enrolled to complete the intervention (i.e., user testing and single-arm pilot participants).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Phase 1 Part 2: Patient User Testing (Months 6-12) and Phase 2: Single-Arm Pilot (Months 12-23)
Number analyzed (Participants) | 37
score on a scale
  0 weeks | 6.05 (2.17)
  12 weeks | 6.88 (1.82)
  16 weeks | 6.90 (1.91)
Statistical Analysis 1: Comparison: Phase 1 Part 2: Patient User Testing (Months 6-12) and Phase 2: Single-Arm Pilot (Months 12-23); 0 to 12 weeks; Test type: Other; Cohen's d effect size = -0.34, 95% CI 2-sided [-0.70 to 0.03]
Statistical Analysis 2: Comparison: Phase 1 Part 2: Patient User Testing (Months 6-12) and Phase 2: Single-Arm Pilot (Months 12-23); 0 to 16 weeks; Test type: Other; Cohen's d effect size = -0.47, 95% CI 2-sided [-0.85 to -0.09]

ADVERSE EVENTS:
Time Frame: Phase 1 Part 1 (Focus Group Patients and Providers): Consent/Enrollment to Completion of One-Time, 60-Minute Telehealth Focus Group, approximately 1-4 weeks. Phase 1 Part 2 (User Testing) and Phase 2 (Single-Arm Pilot): Consent/Enrollment to Completion of 1-Month Post-Treatment Assessment (A3), an average of 16 weeks.
Groups:
- Phase 1 Part 1: Focus Group Patients and Providers (Months 0-6): Patients with hematologic cancer and hematology-oncology providers that consented and enrolled to complete a one-time, 60-minute, telehealth focus group.
- Phase 1 Part 2: Patient User Testing (Months 6-12) and Phase 2: Single-Arm Pilot (Months 12-23): Mindfulness-Based Therapy for Insomnia with Cognitive-Behavioral Symptom Coping Skills (MBTI+)
  The MBTI+ intervention will train participants in mindfulness-based sleep strategies and behavioral symptom management techniques. The MBTI+ intervention will consist of 6 weekly sessions that will last between 60 and 75 minutes.
  Mindfulness-Based Therapy for Insomnia with Cognitive-Behavioral Symptom Coping Skills: Mindfulness-based sleep strategies and cognitive-behavioral symptom coping skills.
Arm/Group | Phase 1 Part 1: Focus Group Patients and Providers (Months 0-6) | Phase 1 Part 2: Patient User Testing (Months 6-12) and Phase 2: Single-Arm Pilot (Months 12-23)
All-Cause Mortality (participants affected / at risk) | 0/20 | 1/37
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/37
Other Adverse Events (participants affected / at risk) | 0/20 | 0/37

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-05-10): https://cdn.clinicaltrials.gov/large-docs/56/NCT04736056/Prot_SAP_001.pdf
  • Informed Consent Form (2023-02-01): https://cdn.clinicaltrials.gov/large-docs/56/NCT04736056/ICF_000.pdf